CLINICAL TRIAL: NCT03245801
Title: The Canadian Alliance of Pediatric Rheumatology Investigators National Juvenile Idiopathic Arthritis Registry
Brief Title: CAPRI National Juvenile Idiopathic Arthritis Registry
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); The Hospital for Sick Children (Other); IWK Health Centre (Other); London Health Sciences Centre (Other); Royal University Hospital Foundation (Other); University of Manitoba (Other); University of Calgary (Other); Alberta Children's Hospital (Other); Memorial University of Newfoundland (Other); McMaster University (Other); McMaster Children's Hospital (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Université de Montréal (Other); Laval University (Other)
Responsible Party: Principal Investigator, Jaime Guzman, Clinical Associate Professor, University of British Columbia
Other Study IDs: H16-00309; UBC Number: F15-01938 (Other Grant/Funding Number: Arthritis Society)
Record Dates: First submitted 2017-07-17; First posted 2017-08-10 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: Juvenile idiopathic arthritis; Canada; Registry; Clinical outcomes; Adverse events; CAPRI
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) is a disorder of unknown cause characterized by chronic inflammation of the joints and other organs. It affects about 1 in a 1000 Canadian children and if untreated it can produce lifelong disability. The Canadian Alliance of Pediatric Rheumatology Investigators (CAPRI) includes most pediatric rheumatologists in Canada. They have successfully collaborated for the past 20 years producing groundbreaking research on the modern course and outcomes of JIA. The CAPRI JIA Registry is an ongoing universal registry of Canadian children with JIA that collects longitudinal data on disease course, outcomes and adverse events to inform healthcare decisions and to gain new insights into the disease and its treatment.

DETAILED DESCRIPTION:
1. BACKGROUND JIA includes all chronic arthritis of unknown cause starting before the age of 16. JIA is the most common rheumatic disease of childhood, affecting approximately 1 in 1,000 Canadian children. Despite trends to more favorable outcomes, JIA continues to have disabling sequelae that reduce mobility, quality of life and future productivity, affecting the child, their families and society as a whole. After a diagnosis of JIA, families have many questions about the prognosis of their child, treatments that may be required and their potential side-effects. Despite numerous studies, our ability to answer these questions remains limited.

   International League of Associations for Rheumatology (ILAR) criteria classify children with JIA into seven categories based on clinical manifestations and laboratory tests. Current practice recommendations propose use of medications tailored according to JIA category or according to treatment groups defined by number of joints affected and features of poor prognosis. In general, initial treatment with intraarticular corticosteroids and nonsteroidal anti-inflammatory drugs (NSAIDs) is recommended for JIA affecting a few joints; while methotrexate and biologic agents are recommended when many joints are affected and for children with features of poor prognosis.

   CAPRI is the collaborative network of all pediatric rheumatology investigators across Canada, with an outstanding track record of successful collaboration in a number of research projects. Since 2005 CAPRI investigators have worked on a project called ReACCH-Out, a team grant funded by the Canadian Institutes of Health Research (CIHR) to study the impact of arthritis on Canadian children. CAPRI developed a robust web-based longitudinal data base and enrolled 1,500 newly diagnosed children with JIA during a five year period. This study has resulted in one of the largest longitudinal JIA cohorts in the world and six published scientific manuscripts to date. Most importantly it has provided essential new answers about disease presentation and short to medium-term prognosis. The initial study was leveraged into two subsequent studies also funded by CIHR: Biologically Based Outcomes Predictors in JIA (BBOP) and Linking Exercise, Activity, and Pathophysiology in Canadian children with Arthritis (LEAP).

   Continuation of this effort with a new registry can illuminate longer term prognosis for JIA patients. The rapidly changing landscape of available therapies necessitates maintenance and extension of the registry to elucidate the changing prognosis in different therapeutic eras, and to enable contemporary prognostic counseling to new patients and their families.

   In April 2015, The Arthritis Society provided an infrastructure award to continue, expand and strengthen a harmonized Canadian registry of patients with JIA, to support pediatric rheumatology research. This award has been enriched with other sources to include assessment of medication adverse events, thus providing the funding that will be used for this CAPRI national JIA registry.
2. GOALS AND PRINCIPLES

The goal of the CAPRI JIA registry is to prospectively collect information on disease course, outcomes and medication adverse events among Canadian children with JIA. The registry will:

1. Provide answers about the expected disease outcomes and the risks of medication adverse events for patients and care providers.
2. Contribute to new insights about JIA and its treatment through yearly updates of registry findings and publication of scientific papers.
3. Allow Canadian researchers to answer their own research questions about JIA.
4. Allow comparison of JIA outcomes and treatments across Canada and with other jurisdictions, in support of quality improvement initiatives.

The registry will operate following five principles:

Universal: all children newly diagnosed with JIA across Canada will be eligible.

Simple: the registry will require minimum training and time to collect information.

High-Quality: the registry will emphasize quality over quantity of data and the quality of data will be continually monitored.

Clinician-centered: the registry will ensure that physicians who follow children with JIA are engaged and see value from their contribution to the registry.

Linkable: the registry will make provisions for future linkages to existing research and healthcare cohorts, to Statistics Canada data and to other databases.

3. METHODS

3.1 Registry oversight

The registry will be managed through CAPRI. A registry committee of CAPRI has been established, with the following responsibilities:

1. Oversight of all registry functions.
2. Report to CAPRI executive.
3. Supervision of the registry coordinator.

The registry committee consists of CAPRI members who volunteer for a 2-year renewable term. The group has elected a chair (Dr. Jaime Guzman) who will be the direct contact for the registry coordinator, organize teleconferences and provide reports to the chair of CAPRI. The registry committee chair will sit on the CAPRI executive committee.

Funding from registry sponsors will come to a central registry account. The registry committee and its chair will be responsible for fund payments, as per agreed CAPRI budget. Financial accounting will be managed by the registry coordinator.

The registry will be subject to the following reporting processes:

1. Annual report to registry sponsors including budget use and progress.
2. Bi-annual report to the CAPRI membership on progress, registry statistics, and budget. A copy of the bi-annual report will be sent to registry sponsors.
3. Annual research output report after the first year of registry operations.
4. Annual update on registry findings to be shared with families and care providers.

3.2 Set up of registry centres All CAPRI centres and pediatric rheumatology practices in Canada are eligible to participate in the registry. Participating sites will designate a registry site director for communication and management purposes. Each site will be responsible for patient enrollment, data entry, and maintenance of appropriate registry records for their site. The registry site director will manage their own site budget, and be required to provide annual budget records.

The registry coordinator will assist each registry site in completing the following steps necessary for set up:

1. Submission of registry protocol for ethics review by the local ethics board and amendments as needed
2. Deciding on the logistics of patient recruitment and registration that best fit with the centre current practices and processes.
3. Deciding on the logistics of data collection that best fit their local practices and processes, including timelines for data submission and locking of the data.
4. Review and agree on the processes for data quality monitoring.

3.3 Patient recruitment and registration At the medical visit where a new diagnosis of JIA is made, the pediatric rheumatologist making the diagnosis will introduce the registry to the patient. The registry site director or delegate will then provide the family with full information about the registry and ask for their written consent. ReACCh-Out and LEAP participants will be asked to re-consent for the registry at their first regular visit.

Registration includes three steps:

1. Review and signing of the consent form
2. Assignment of a unique registry identification number by an automated online system
3. Collection of initial registry data as described below

3.4 Data collection The registry will collect data from the pediatric rheumatologist caring for the child, and from the child and the child's parent or guardian. Data will be collected from the physician and families at registration followed by a minimum set of data at every subsequent clinic visit. Additional data once yearly at a visit close to the anniversary of the diagnosis will be collected from families. All data will be collected at clinic visits and there will be no visits booked specifically for registry purposes.

The primary method of data collection from physicians will be direct entry online using a secure web site located at a Canadian academic centre, via computer or smart phone. The secondary method of data collection will be in paper forms for physicians who prefer that method. Data in paper forms will then be entered online by research assistants.

The primary method of data collection from families will be in paper forms. The answers will be verified by research assistants and then entered online. The secondary method of data collection will be direct entry online for centres where existing infrastructure allows for direct entry by families at the time of the visit.

3.5 Protection of privacy and confidentiality All data collected will be handled in accordance with federal and provincial personal information legislation. Information that would allow identification of a child, such as name, date of birth and address will only be collected in the consent form. This information will be separate from registry information and will not be available in any online system. All subsequent data collection will have no personal identifying information, only the registry identification number.

The de-identified registry information will be stored online in a dedicated RedCap server at a Canadian academic centre that complies with all encryption and audit regulatory requirements. As this is an ongoing registry de-identified electronic records will be kept indefinitely in the secure servers. There is a possibility in the future to have international collaborations to help with data analysis. In this case, data sent outside of Canada will not contain any personal identifying information and will be strictly de-identified.

Any de-identified paper records used during the process of entering information in the registry will be kept under locked storage for ten years and then destroyed. They are to be used in case of need for confirmation of the veracity of the data for scientific publication purposes.

3.6 Data quality monitoring

The continuous monitoring of data quality is an essential function of the registry and the major responsibility of the registry coordinator. The registry committee and its chair bear final accountability for the quality of the data entered in the registry. The following four complementary methods will ensure the data contained in the registry is complete and of the highest possible quality:

1. Quality control during data entry: Defines the automatic quality controls set up as part of data entry for each questionnaire or form.
2. Daily quality control by registry coordinator: Defines the daily activities of the registry coordinator to monitor data quality and actions to follow through on issues identified.
3. Quality control at periodic centre audits: Defines indications for quality audits, their periodicity and how their results are assessed and followed through.
4. Monthly update on quality control to registry chair: defines the components of the monthly quality update, how it is prepared and how it is assessed by the chair.

3.7 Access to data To assist healthcare provision: Patients and their physicians will have access to their data to obtain estimates of expected outcomes and risks of side effects based on analyses of registry data.

To answer research questions: CAPRI and non-CAPRI researchers may request access to registry data to answer research questions.

To assist planning and program development: Healthcare organizations, registry sponsors, health authorities and ministries of health services, may request access to summary statistics or de-identified group data for use in knowledge translation activities or to assist in their planning of programs and delivery of care.

ELIGIBILITY:
Inclusion Criteria:

1. All patients newly diagnosed with JIA within the last 3 months
2. All patients who participated in the original ReACCh-Out study
3. LEAP study patients from 'newly diagnosed' and 'ReACCh-Out' cohorts who have completed their two year follow up in LEAP

Exclusion Criteria:

1. Patients with an unconfirmed JIA diagnosis
2. Patients diagnosed with JIA more than 3 months prior to the clinic visit, who were not followed in LEAP and /or ReACCh-Out studies.
3. If the family as a whole is unable to answer questionnaires in English or French

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric rheumatology clinic patients at study sites
Sampling Method: Non-Probability Sample
Enrollment: 1238 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Children with Clinical inactive disease | At one year
  This is an accepted validated composite measure requiring all of the following: No active joints, no extra-articular manifestations, a physician global assessment of disease activity of less than 1, morning stiffness of 15 min or less, and normal inflammatory markers (ESR or CRP).

SECONDARY OUTCOMES:
Juvenile Arthritis Disease Activity Score | One year
  This is an accepted validated measure composed of the sum of physician global assessment, parent global assessment and up to 10 active joints.
Pain intensity | One year
  Severity of arthritis pain in the last week, from 0 to 10
Juvenile Arthritis Quality of Life Questionnaire | One year
  Composite measure of quality of life with total of 72 items, score from 1 (best) to 7 (worst) quality of life.
Childhood Health Assessment Questionnaire Disability Index | One year
  Composite measure of functional disability, score from 0 (no disability) to 3 (severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Guzman, MD, FRCPC, Study Chair — University of British Columbia; Adam Huber, MD, Principal Investigator — IIWK Health Centre, Halifax, Nova Scotia, Canada; Ciaran Duffy, MD, Principal Investigator — Children's Hospital of Eastern Ontario, Ottawa, Ontario; Gaëlle Chédeville, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Heinrike Schmeling, MD, Principal Investigator — Alberta Children's Hospital; Linda Hiraki, MD,FRCPC,MS, Principal Investigator — Hospital for Sick Children (SickKids); Heinrike Schmeling, MD, Principal Investigator — University of Calgary / Alberta Children's Hospital; Susanne Benseler, MD, PhD, Principal Investigator — University of Calgary / Alberta Children's Hospital; Marinka Twilt, MD MSCE PhD, Principal Investigator — University of Calgary / Alberta Children's Hospital
Locations (15):
- Canada (15):
  - University of Calgary / Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - University of Manitoba/Children's hospital research institute, Winnipeg, Manitoba
  - Memorial University/Janeway Childrens Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador, Canada
  - IIWK Health Centre, Halifax, Nova Scotia
  - McMaster University/McMaster Children's Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Université de Montréal, Montreal, Quebec
  - University of Sherbrooke, Sherbrooke, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - CHU Québec - Universite Laval, Québec

IPD SHARING:
Plan to Share IPD: Yes
CAPRI researchers who seek to use de-identified registry data to answer research questions not contemplated in this protocol will apply through the CAPRI Scientific Protocol Evaluation Committee (SPEC) process and produce proof of ethics board approval before release of data. Registry site directors will have access to their local data for smaller local research projects. Provision of information regarding project title, aim, and any ensuing publication will be required so that a complete record of research projects can be maintained. Non-CAPRI researchers who seek access to registry data must have a research team that includes at least one CAPRI member and apply for use through the CAPRI SPEC. Proof of ethics board approval will be required before release of data. All research abstracts, presentations and publications using registry data must acknowledge registry sponsors.The registry committee and CAPRI executive will determine data access recovery fees.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Ongoing, as long as the Registry is in operation.
Access Criteria: Non-CAPRI researchers who seek access to registry data must have a research team that includes at least one CAPRI member and apply for use through the CAPRI SPEC. Proof of ethics board approval will be required before release of data.

REFERENCES:
- [Background] Petty RE, Southwood TR, Manners P, Baum J, Glass DN, Goldenberg J, He X, Maldonado-Cocco J, Orozco-Alcala J, Prieur AM, Suarez-Almazor ME, Woo P; International League of Associations for Rheumatology. International League of Associations for Rheumatology classification of juvenile idiopathic arthritis: second revision, Edmonton, 2001. J Rheumatol. 2004 Feb;31(2):390-2. No abstract available. PMID 14760812
- [Background] Shiff NJ, Lix LM, Oen K, Joseph L, Duffy C, Stringer E, Tucker LB, Svenson LW, Belisle P, Bernatsky S. Chronic inflammatory arthritis prevalence estimates for children and adolescents in three Canadian provinces. Rheumatol Int. 2015 Feb;35(2):345-50. doi: 10.1007/s00296-014-3085-0. Epub 2014 Jul 15. PMID 25023756
- [Background] Oen K. Long-term outcomes and predictors of outcomes for patients with juvenile idiopathic arthritis. Best Pract Res Clin Rheumatol. 2002 Jul;16(3):347-60. PMID 12387804
- [Background] Ravelli A, Martini A. Early predictors of outcome in juvenile idiopathic arthritis. Clin Exp Rheumatol. 2003 Sep-Oct;21(5 Suppl 31):S89-93. PMID 14969057
- [Background] Adib N, Silman A, Thomson W. Outcome following onset of juvenile idiopathic inflammatory arthritis: I. frequency of different outcomes. Rheumatology (Oxford). 2005 Aug;44(8):995-1001. doi: 10.1093/rheumatology/keh620. Epub 2005 Apr 12. PMID 15827045
- [Background] Dueckers G, Guellac N, Arbogast M, Dannecker G, Foeldvari I, Frosch M, Ganser G, Heiligenhaus A, Horneff G, Illhardt A, Kopp I, Krauspe R, Markus B, Michels H, Schneider M, Singendonk W, Sitter H, Spamer M, Wagner N, Niehues T. Evidence and consensus based GKJR guidelines for the treatment of juvenile idiopathic arthritis. Clin Immunol. 2012 Feb;142(2):176-93. doi: 10.1016/j.clim.2011.10.003. Epub 2011 Oct 26. PMID 22154868
- [Background] Beukelman T, Patkar NM, Saag KG, Tolleson-Rinehart S, Cron RQ, DeWitt EM, Ilowite NT, Kimura Y, Laxer RM, Lovell DJ, Martini A, Rabinovich CE, Ruperto N. 2011 American College of Rheumatology recommendations for the treatment of juvenile idiopathic arthritis: initiation and safety monitoring of therapeutic agents for the treatment of arthritis and systemic features. Arthritis Care Res (Hoboken). 2011 Apr;63(4):465-82. doi: 10.1002/acr.20460. PMID 21452260
- [Background] Oen K, Duffy CM, Tse SM, Ramsey S, Ellsworth J, Chedeville G, Chetaille AL, Saint-Cyr C, Cabral DA, Spiegel LR, Schneider R, Lang B, Huber AM, Dancey P, Silverman E, Rosenberg AM, Cameron B, Johnson N, Dorval J, Scuccimarri R, Campillo S, Petty RE, Duffy KN, Boire G, Haddad E, Houghton K, Laxer R, Turvey SE, Miettunen P, Gross K, Guzman J, Benseler S, Feldman BM, Espinosa V, Yeung RS, Tucker L. Early outcomes and improvement of patients with juvenile idiopathic arthritis enrolled in a Canadian multicenter inception cohort. Arthritis Care Res (Hoboken). 2010 Apr;62(4):527-36. doi: 10.1002/acr.20044. PMID 20391508
- [Background] Guzman J, Oen K, Huber AM, Watanabe Duffy K, Boire G, Shiff N, Berard RA, Levy DM, Stringer E, Scuccimarri R, Morishita K, Johnson N, Cabral DA, Rosenberg AM, Larche M, Dancey P, Petty RE, Laxer RM, Silverman E, Miettunen P, Chetaille AL, Haddad E, Houghton K, Spiegel L, Turvey SE, Schmeling H, Lang B, Ellsworth J, Ramsey SE, Bruns A, Roth J, Campillo S, Benseler S, Chedeville G, Schneider R, Tse SM, Bolaria R, Gross K, Feldman B, Feldman D, Cameron B, Jurencak R, Dorval J, LeBlanc C, St Cyr C, Gibbon M, Yeung RS, Duffy CM, Tucker LB; ReACCh-Out investigators. The risk and nature of flares in juvenile idiopathic arthritis: results from the ReACCh-Out cohort. Ann Rheum Dis. 2016 Jun;75(6):1092-8. doi: 10.1136/annrheumdis-2014-207164. Epub 2015 May 18. PMID 25985972
- [Background] Guzman J, Oen K, Tucker LB, Huber AM, Shiff N, Boire G, Scuccimarri R, Berard R, Tse SM, Morishita K, Stringer E, Johnson N, Levy DM, Duffy KW, Cabral DA, Rosenberg AM, Larche M, Dancey P, Petty RE, Laxer RM, Silverman E, Miettunen P, Chetaille AL, Haddad E, Houghton K, Spiegel L, Turvey SE, Schmeling H, Lang B, Ellsworth J, Ramsey S, Bruns A, Campillo S, Benseler S, Chedeville G, Schneider R, Yeung R, Duffy CM; ReACCh-Out investigators. The outcomes of juvenile idiopathic arthritis in children managed with contemporary treatments: results from the ReACCh-Out cohort. Ann Rheum Dis. 2015 Oct;74(10):1854-60. doi: 10.1136/annrheumdis-2014-205372. Epub 2014 May 19. PMID 24842571
- [Background] Shiff NJ, Tucker LB, Guzman J, Oen K, Yeung RS, Duffy CM. Factors associated with a longer time to access pediatric rheumatologists in Canadian children with juvenile idiopathic arthritis. J Rheumatol. 2010 Nov;37(11):2415-21. doi: 10.3899/jrheum.100083. Epub 2010 Aug 17. PMID 20716664
- [Background] Oen K, Tucker L, Huber AM, Miettunen P, Scuccimarri R, Campillo S, Cabral DA, Feldman BM, Tse S, Chedeville G, Spiegel L, Schneider R, Lang B, Ellsworth J, Ramsey S, Dancey P, Silverman E, Chetaille AL, Cameron B, Johnson N, Dorval J, Petty RE, Duffy KW, Boire G, Haddad E, Houghton K, Saint-Cyr C, Turvey SE, Benseler S, Cheang M, Yeung RS, Duffy CM. Predictors of early inactive disease in a juvenile idiopathic arthritis cohort: results of a Canadian multicenter, prospective inception cohort study. Arthritis Rheum. 2009 Aug 15;61(8):1077-86. doi: 10.1002/art.24539. PMID 19644903
- See also: Juvenile idiopathic arthritis — https://ghr.nlm.nih.gov/condition/juvenile-idiopathic-arthritis